CLINICAL TRIAL: NCT03610997
Title: Photorefractive Keratectomy for Anisometropic and Isoametropic Amblyopia in Children Refractory to Conventional Treatment
Brief Title: Photorefractive Keratectomy for Severe Anisometropia and Isoametropia Associated With Amblyopia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants no longer receiving intervention
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Evelyn Paysse, Professor of Ophthalmology and Pediatrics, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-6604
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Anisometropia; Hyperopia; High Myopia; Amblyopia Isometropic; Amblyopia Bilateral; High Astigmatism
MeSH Terms: conditions — Anisometropia; Hyperopia | interventions — Photorefractive Keratectomy

STUDY DESIGN:
Intervention Model Description: Photorefractive Keratectomy
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Photorefractive keratectomy (Other): The children will undergo PRK in the affected eye(s) using previously derived formulas for PRK.
  Interventions: Procedure: Photorefractive keratectomy

INTERVENTIONS:
Procedure: Photorefractive keratectomy

SUMMARY:
Photorefractive keratectomy (PRK) with excimer laser has been used successfully to treat myopia, hyperopia, and astigmatism in adults for over 35 years. Children with high refractive errors that go untreated will develop severe amblyopia. PRK can normalize high refractive errors and potentially improve the visual acuity in affected children. The purpose of this study is to investigate whether children with high anisometropia or isoametropia with amblyopia that are nonresponsive to standard therapy and receive PRK develop better longterm visual acuity.

DETAILED DESCRIPTION:
Anisometropia is a condition in which one eye has a significantly different refractive error from the other and commonly leads to the development of refractive amblyopia in the affected eye. High isoametropia is the condition in which both eyes have high refractive error and commonly leads to bilateral refractive amblyopia if untreated. Amblyopia is the condition in which vision does not develop fully in the brain due to disuse or misuse of one or both eyes. Typically, in high anisometropia, a contact lens in the eye with the stronger refractive error and/or glasses must be used to correct the refractive error. Commonly, infants and children with this condition refuse to wear the contact lens or glasses because the other eye sees normally. There are other problems in treating high anisometropia with glasses. One is aniseikonia, the condition of image size disparity between the two eyes. This causes difficulty for the brain of the affected person to fuse the images from the two eyes because the image from one eye is much larger than that from the other eye. This results in asthenopia (eye fatigue) and sometimes even diplopia. If the anisometropia is severe, significant amblyopia will result in the eye with the stronger refractive error and, if not treated at an early age, permanent and potentially severe vision loss will result.

In high isoametropia, contact lenses or glasses must likewise be used in order for normal vision to develop. Most children with isoametropia will wear glasses well because they cannot see well without them. By contrast, children with developmental delays, chromosomal abnormalities, autism, or attention deficit hyperactivity disorder and high isoametropia very commonly will not wear the needed refractive correction due to strong tactile aversion to anything touching their face or head. If the refractive error is high, significant bilateral (isoametropic) amblyopia will result and, if not treated at an early age, permanent and potentially severe vision loss will result.

PRK can normalize high refractive errors and potentially reduce or eliminate the amblyopia in affected children. The purpose of this study is to investigate whether children with high anisometropia or isoametropia with amblyopia that are nonresponsive to standard therapy and receive PRK develop better longterm visual acuity. Secondary outcomes are stability of refractive correction, and corneal health.

ELIGIBILITY:
Inclusion Criteria:.

* Children aged 2 to 17 with significant anisometropia or isoametropia and amblyopia that have failed traditional treatment for at least 6 months.
* Anisometropic group:
* The anisometropia must be at least 3.00 diopters.
* The amblyopic eye best corrected visual acuity must be at least 2 lines worse than the fellow eye in verbal children
* Isoametropic group
* Myopia must be at least -4.00 diopters in both eyes
* Hyperopia must be at least +4.00 diopters in both eyes
* Astigmatism must be at least +2.50 diopters in both eyes.

Exclusion Criteria:

* History of significant corneal abnormality that, in the investigator's opinion, may limit visual rehabilitation.
* History of known collagen disorder
* History of known corneal ectasia
* History of previous herpes simplex keratitis
* Corneal thickness of less than 450u

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 10 years
  Snellen equivalent

SECONDARY OUTCOMES:
Refractive error | 10 years
  cycloplegic refraction
Corneal clarity | 10 years
  slit lamp exam

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Paysse, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No